CLINICAL TRIAL: NCT00520663
Title: An Open-label Study to Determine the Excretion, Balance and Pharmacokinetics of SB649868 After a Single Oral Administration of 14C-SB649868 in Healthy Volunteers
Brief Title: Radiolabel Study In Healthy Volunteers For Insomnia-Targeting Drug
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXS109139
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Distribution,; SB-649868,; Healthy,; Excretion,; Sleep disturbances; Volunteer,; Metabolism,; Absorption,
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias | interventions — N-((1-((5-(4-fluorophenyl)-2-methyl-4-thiazolyl)carbonyl)-2-piperidinyl)methyl)-4-benzofurancarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy male subjects (Experimental): Each subject will receive a single oral dose of 14C-SB649868 (containing approximately 70 microcuries of radiocarbon and 30 milligrams of SB649868).
  Interventions: Drug: 14C-SB649868

INTERVENTIONS:
Drug: 14C-SB649868 — SB-649868 will be provided as powder in a bottle which will be reconstituted into a solution prior to dosing via a hard gelatin capsule. Each subject will receive one unit dose of SB-649868 30 milligram reconstituted powder presented in a size 00 capsule once. The capsule will be swallowed with 160 milliliters of water.

SUMMARY:
The purpose of this study is to define the absorption, breakdown and excretion of a single dose of radiolabelled SB-649868 and its breakdown products by measuring their concentration in blood, urine and faeces over a 7-10 day period. "Radiolabelled" means that the test drug has a radioactive component to help us track the drug. The safety and tolerability of the test drug will also be assessed.

ELIGIBILITY:
Inclusion criteria:

* Healthy males, aged 30-55 years inclusive.
* Body weight more or equal to 50kg with a BMI (body mass index) between 18.5-29.9kg/m2 inclusive.
* Healthy as based on a medical evaluation consisting of medical history, physical examination, lab tests on blood and urine and cardiovascular monitoring.

LH, FSH and testosterone hormones must be within normal reference range.

Exclusion criteria:

* Positive urine drug screen or alcohol breath test at screening visit.
* Average weekly alcohol intake of more than 21 units or average daily intake of more than 3 units.
* Grapefruit or grapefruit juice intake 7 days before dosing and until the last blood sample is taken.
* Any subject who is not prepared to eat standard meals in the clinic or is a vegetarian.
* Participated in a clinical trial for a new drug within 30 days or 5 half-lives or twice the duration of that drugs effect before the dosing day for this study.
* Exposure to 4 new drugs in clinical trials within the last 12 months before dosing in this study.
* Use of any medications (prescribed or non-prescribed including vitamins and herbal supplements) within 7 days before dosing in this study.
* Participation in this study would result in the subject donating more than 500ml in a 56 day period.
* Regular use of tobacco or nicotine-containing products within 6 months of screening.
* Unwillingness to abstain from sexual intercourse with pregnant or lactating women from dosing until 84 days after.
* Unwillingness to use contraception and have female partner use contraception if she could become pregnant for 84 days after dosing.
* Unwillingness to abstain from strenuous physical activity for 48 hours before screening and in the 72 hours before and 48 hours after the treatment period.
* Administration of radiolabelled substances or exposure to significant radiation (eg serial X-rays or CT scans, barium meal etc)within the past 12 months from screening.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2007-06-08 (Actual); Primary Completion 2007-08-10 (Actual); Study Completion 2007-08-10 (Actual)

PRIMARY OUTCOMES:
Excretion of SB649868 by measuring radioactivity in urine and faeces | over 7-10 days.
Plasma levels of SB-649868 by measuring drug levels and radioactivity in plasma. Plasma, urine,faeces samples to study the metabolites of SB649868. | over 4 days

SECONDARY OUTCOMES:
Safety and tolerability of 14C-SB649868 by adverse event monitoring, lab samples and cardiovascular monitoring. | over the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tranent, West Lothian, United Kingdom

REFERENCES:
- See also: Results for study 109139 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/OXS109139?search=study&search_terms=OXS109139#rs